CLINICAL TRIAL: NCT00043693
Title: Family Intervention for SMI and Substance Use Disorder
Brief Title: Family Intervention for Mental Illness and Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH062629 (NIH); R01MH062629 (NIH); DSIR SE-CE
Record Dates: First submitted 2002-08-12; First posted 2002-08-15 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia; Bipolar Disorder; Substance-related Disorders
Keywords: Psychotic Disorders; Schizoaffective Disorder; Substance Abuse
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Substance-Related Disorders; Psychotic Disorders | interventions — mica

ARMS (2):
- 1 (Experimental): Participants will undergo the Family Intervention for Dual Diagnosis (FIDD) program.
  Interventions: Behavioral: Family Intervention for Dual Diagnosis
- 2 (Active Comparator): Participants will be placed in a family psychoeducation program.
  Interventions: Behavioral: Family psychoeducation program

INTERVENTIONS:
Behavioral: Family Intervention for Dual Diagnosis — The family intervention for dual diagnosis program lasts for up to 3 years and includes both single and multiple-family group formats.
  Arms: 1
Behavioral: Family psychoeducation program — The family psychoeducation program consists of 6 weekly sessions.
  Arms: 2

SUMMARY:
This study will evaluate a family intervention program for individuals with bipolar disorder, schizophrenia, or schizoaffective disorder and co-occurring substance use disorders.

DETAILED DESCRIPTION:
Substance use disorder (SUD) in persons with severe mental illness may worsen the course of psychiatric illness. The loss of family support for individuals with mental illness is a major contributing factor to housing instability, homelessness, and other problems. Despite progress toward integrating mental health and substance abuse services, interventions that improve the course of mental illness while helping the families of the mentally ill are not currently available. Enhancing skills for coping with mental illness may be an effective strategy for treating SUD, decreasing caregiver burden, and improving the long-term outcomes for people with mental illness.

Patients and their families are randomly assigned to either the Family Intervention for Dual Diagnosis (FIDD) program or family psychoeducation. The FIDD program lasts for up to 3 years and includes both single and multiple-family group formats. The family psychoeducation program consists of 6 weekly sessions. Routine assessments are conducted on all patients, and relatives are evaluated on a wide range of outcomes, including substance abuse, hospitalizations, psychiatric symptoms, legal problems, aggression, housing and homelessness, family burden, social support, and quality of life. To determine the effectiveness of the FIDD program, knowledge of mental illness and problem-solving skills are assessed in the families following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have schizophrenia, schizoaffective disorder, or bipolar disorder
* Have a current substance use disorder (within the past 6 months)
* Are willing to have at least 4 hours of contact per week with family members or significant others
* Plan to remain in the community
* Have family members or significant others who consent to participate in the study and plan to remain in the community

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2002-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Alcohol use scale-revised | Measured at baseline, during treatment, and post-treatment
Drug use scale-revised | Measured at baseline, during treatment, and post-treatment
Substance abuse treatment scale | Measured at baseline, during treatment, and post-treatment
Timeline followback calandar | Measured at baseline, during treatment, and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kim T. Mueser, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Shirley Glynn, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Pacific Clinics El Camino, Santa Fe Springs, California
  - North Suffolk Mental Health Association, Chelsea, Massachusetts

REFERENCES:
- [Background] Mueser KT, Fox L. A family intervention program for dual disorders. Community Ment Health J. 2002 Jun;38(3):253-70. doi: 10.1023/a:1015271908765. PMID 12046678